CLINICAL TRIAL: NCT05479591
Title: Glycaemic Control and Management in Adult Type 2 Diabetes Patients Previously Treated With Premix Insulins and Initiating Treatment With IDegLira in Routine Clinical Practice in Croatia: A 36-week Single Arm, Prospective, Multi-centre, Non-interventional Study
Brief Title: A Research Study Looking at Blood Sugar Control in People With Type 2 Diabetes Previously Treated With Premix Insulin and Initiating Treatment With Insulin Degludec/Liraglutide (IDegLira) in Local Clinical Practice in Croatia
Acronym: GLIDE
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9068-4972; U1111-1271-8967 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — IDegLira; Xultophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with type 2 diabetes (T2D): Participants with T2D previously treated with premix insulin for at least 12 weeks (3 months) based on local clinical guidelines will initiate treatment with IDegLira at the treating physician's discretion according to the approved IDegLira label in Croatia.
  Interventions: Drug: IDegLira

INTERVENTIONS:
Drug: IDegLira — Participants will be treated with IDegLira at the treating physician's discretion according to the approved IDegLira label in Croatia and independent from the decision to include the participant in the study.
  Other Names: Xultophy

SUMMARY:
The purpose of this study is to look at the blood sugar control in participants with type 2 diabetes previously treated with premix insulins and initiating treatment with IDegLira. Participants will get IDegLira as prescribed by study doctor regardless of participant's decision to participate in the study. Decision to initiate treatment with IDegLira will be made by study doctor independent from the study. The study will last for about 36 weeks. Participants will be asked questions about their health and diabetes treatment and lab tests as part of their normal doctor's appointment.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female patients aged greater than or equal to (>=) 18 years at the time of signing informed consent.
* Patients diagnosed with T2D and receiving treatment with premix insulin for at least 12 weeks (3 months) based on local clinical guidelines.
* Switched to treatment with IDegLira from previous treatment of premix insulins. The decision to initiate treatment with IDegLira must be independently from the decision to enrol in the study.
* Available and documented HbA1c collected within 12 weeks prior to initiation of IDegLira.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Participation in any other T2D clinical trial of an approved or non-approved investigational medicinal product within 30 days prior to initiation of IDegLira.
* Previous treatment with IDegLira.
* Patients diagnosed with Type 1 diabetes mellitus.
* Female who is known to be pregnant, breastfeeding or intends to become pregnant during the conduct of the study.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Known or suspected hypersensitivity to the active substance or to any of the excipients as specified in the IDegLira label in Croatia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Type 2 Diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Glycated Haemoglobin A1c (HbA1c) | From baseline to end of study (week 36 ± 6 weeks)
  Measured in percentage (%) point.

SECONDARY OUTCOMES:
Number of participants with HbA1c less than (<) 7.0% | At end of study (week 36 ± 6 weeks)
  Number of participants having Yes/No.
Starting dose of IDegLira | At baseline
  Measured in dose steps/day.
Dose of IDegLira at end of study | At end of study (week 36 ± 6 weeks)
  Measured in dose steps/day.
Change in body weight | From baseline to end of study (week 36 ± 6 weeks)
  Measured in kilograms (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com